CLINICAL TRIAL: NCT04070001
Title: Comparison of the Effects of Ibuprofen and Low-Level Laser Therapy on Orthodontic Pain By Means of Interleukin 1-Beta and Substance P Levels in the Gingival Crevicular Fluid
Brief Title: The Effects of Ibuprofen and Laser on Orthodontic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yeşim KAYA (Other)
Responsible Party: Sponsor-Investigator, Yeşim KAYA, Assistant professor, Yuzuncu Yil University
Organization: Yuzuncu Yil University (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: 26.07.2017/04
Record Dates: First submitted 2019-08-22; First posted 2019-08-28 (Actual); Last update posted 2019-08-29 (Actual); Status verified 2019-08

CONDITIONS: Crowding, Tooth
Keywords: Pain; Elastomeric separator; Laser; Ibuprofen; Gingival crevicular fluid
MeSH Terms: conditions — Malocclusion; Pain | interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Ibuprofen group (Active Comparator): Ibuprofen group received 1-dose 400-mg Ibuprofen 1 hour before elastomeric separator placement
  Interventions: Drug: 400 Mg Ibuprofen
- Laser group (Active Comparator): Laser groups received a single irradiation of low-level laser immediately after elastomeric separator placement.
  Interventions: Device: laser application
- Control group (Placebo Comparator): Control group received placebo lactose tablets 1 hour before elastomeric separator placement.
  Interventions: Other: placebo tablets

INTERVENTIONS:
Drug: 400 Mg Ibuprofen — 1-dose 400-mg ibuprofen 1-hour before elastomeric separator placement
  Arms: Ibuprofen group
Device: laser application — A single irradiation of laser after elastomeric separator placement
  Arms: Laser group
Other: placebo tablets — Placebo lactose tablets 1-hour before elastomeric separator placement
  Arms: Control group

SUMMARY:
Early orthodontic pain is usually caused by the insertion of elastomeric separators to the mesial and distal of the tooth to be banded in order to create adequate space for proper placement. Recent studies have demonstrated that the pain reaches its peak at 24 hours and then gradually decreases within 7 days The intensity of this pain is sometimes perceived as extremely high to cause a significant number of patients to discontinue the treatment.

Nonsteroidal anti-inflammatory drugs, which block the prostaglandin synthesis through inhibiting the cyclooxygenase activity, is one of the most common methods used to manage the orthodontic pain. It has been reported that these drugs decrease the orthodontic tooth movement rate, in addition to many systemic side effects such as gastric and duodenal ulceration, coagulation disorders, congestive heart problems and allergic effect.

The application of low-level laser therapy (LLLT) also reported being efficient in accelerating orthodontic tooth movement and in alleviating orthodontic pain without any apparent side effects. LLLT is thought to reduce the pain by increasing the local blood flow, inhibiting the secretion of inflammatory substances, inducing the release of neurotransmitters, altering the conduction and excitation of peripheral nerves and stimulating the endorphins release. On the other hand, literature review on the effectiveness of LLLT in alleviating orthodontic pain observed after elastomeric separator placement (ESP) exhibited conflicting results. While LLLT was found to be effective in some studies, the others refuted its effectiveness.

When studies on alleviating orthodontic pain observed after ESP were reviewed, it was determined that the effects of many drugs and LLLT were evaluated subjectively by VAS. Furthermore, only in one study, the effects of ibuprofen and LLLT were compared using PGE2 levels in GCF and VAS. Based on that, this study was aimed to compare the effects of ibuprofen and LLLT in alleviating orthodontic pain observed after ESP through IL-1β and SP levels in GCF and VAS.

DETAILED DESCRIPTION:
Pain is defined as a sophisticated experience that includes sensations evoked by, and reactions to noxious stimuli. During the different phase of orthodontic treatment, pain is developed in response to the tension and pressure zones generated in the periodontal ligament following the force application. This leads to the secretion of inflammatory mediators such as histamine, serotonin, dopamine, glycine, cytokines, leukotrienes, prostaglandins and substance P that stimulate free nerve endings resulting in the perception of pain.

Early orthodontic pain is usually caused by the insertion of elastomeric separators to the mesial and distal of the tooth to be banded in order to create adequate space for proper placement. Recent studies have demonstrated that the pain reaches its peak at 24 hours and then gradually decreases within 7 days. The intensity of this pain is sometimes perceived as extremely high to cause a significant number of patients to discontinue the treatment.

Nonsteroidal anti-inflammatory drugs, which block the prostaglandin synthesis through inhibiting the cyclooxygenase activity, is one of the most common methods used to manage the orthodontic pain. It has been reported that these drugs decrease the orthodontic tooth movement rate, in addition to many systemic side effects such as gastric and duodenal ulceration, coagulation disorders, congestive heart problems and allergic effect.

The application of low-level laser therapy (LLLT) also reported being efficient in accelerating orthodontic tooth movement and in alleviating orthodontic pain without any apparent side effects. LLLT is thought to reduce the pain by increasing the local blood flow, inhibiting the secretion of inflammatory substances, inducing the release of neurotransmitters, altering the conduction and excitation of peripheral nerves and stimulating the endorphins release. On the other hand, literature review on the effectiveness of LLLT in alleviating orthodontic pain observed after elastomeric separator placement (ESP) exhibited conflicting results. While LLLT was found to be effective in some studies, the others refuted its effectiveness.

The intensity of orthodontic pain was evaluated either subjectively by visual analog scale (VAS) or objectively by chemical analysis of gingival crevicular fluid (GCF), in previous studies. The analysis of GCF is a useful and non-invasive method for detecting the biochemical mediators released during tooth movement with reasonable sensitivity. In GCF, pro-inflammatory mediators such as interleukin 1-beta (IL-1β) and prostaglandin E2 (PGE2) and neuropeptides such as Substance P (SP) have been related separately to pain. When studies on alleviating orthodontic pain observed after ESP were reviewed, it was determined that the effects of many drugs and LLLT were evaluated subjectively by VAS. Furthermore, only in one study, the effects of ibuprofen and LLLT were compared using PGE2 levels in GCF and VAS. Based on that, this study was aimed to compare the effects of ibuprofen and LLLT in alleviating orthodontic pain observed after ESP through IL-1β and SP levels in GCF and VAS. The null hypothesized was that there was no difference between the effects of ibuprofen and LLLT in orthodontic pain relief.

A total of 60 subjects who referred to the Department of Orthodontics, Faculty of Dentistry at XXXX University between October 2017 and January 2019, were included in this randomized controlled clinical trial. The inclusion criteria were as follows: being older than 18 years of age, requiring ESP at the beginning of orthodontic treatment for banding of maxillary first molars, intact maxillary dentition (exception of third molars), fully erupted maxillary first molars without any treated or not treated apical lesions, tight contacts between the posterior teeth, no pregnancy and lactation, the absence of systemic and periodontal diseases and chronic or neural pains, currently not using analgesics or antibiotics that interfere the pain perception, no contradiction to the use of ibuprofen, the absence of gingival pigmentation where the laser will be applied. The exclusion criteria were: previous orthodontic treatment, falling to complete the questionnaire and to continue to the follow-up appointments.

Sample size calculation Depending on the results of previous studies the standard deviation (σ) was considered as 11 mg/dl in this study. Furthermore, for the 0.05 type I error rate the effect size, and Z values were assumed to be 5 and 1.96, respectively. Based on this information, the sample size was found to be a minimum of 18.6 (≅19) according to the equation of sample size calculation (n=Z2σ2/d2).

Randomization The subjects were randomly assigned to ibuprofen, laser, and control groups using a simple randomization technique. The investigators asked each subject to choose one of the 60 closed envelopes that were equally divided into all groups. The male to female ratio was also equal in each group. An operator outside the study performed the random allocation. Elastomeric separators (3M Unitek, Monrovia, Calif) were inserted by a single investigator (YK) at the mesial and distal interproximal spaces of the maxillary first molars.

Study groups While the ibuprofen group received 400-mg ibuprofen orally 1 hour before ESP, the laser group received a single irradiation of low-level laser immediately after ESP. Likewise, placebo lactose tablets were given orally to the control group 1 hour before ESP. The ibuprofen and placebo lactose tablets were placed in identical capsules in order to blind the subjects and investigator to the treatment group. Subjects were told not to take any other analgesic during the observation period.

Laser parameters and procedure An 810-nm semi-conductor Gallium Aluminum Arsenide (Ga-Al-As) diode laser device (Cheese Diode Laser, Wuhan Gigaa Optronics Technology Co. Ltd., China) with continuous emission mode was used for this study. For each quadrant, a total of 8 doses of laser irradiation (2 J/cm2, 100mW, 10 sn) were applied to the cervical third of the roots. The mesial and distal of the first molars, mesial of the second premolars and distal of the second molars were irradiated from both buccal and palatal sides. During the exposure, the tip held perpendicular and in contact with the mucosa.

Pain assessment Subject's pain intensity was evaluated by means of a questionnaire containing VAS (10-cm horizontal line with the number 0 representing no pain and the number 10 representing the worst pain). While baseline evaluations were made immediately after ESP in the ibuprofen and control groups, it was made after laser application in the laser group. The remaining evaluations were performed at the 2nd and 6th hours, and on the 1st, 3rd, and 7th days. Each subject was asked to mark a vertical line crossing the horizontal line, which best represented the perceived level of pain, on the questionnaire containing the evaluation time points given to them.

Gingival crevicular fluid (GCF) sampling GCF samples were collected from the mesiobuccal and distobuccal gingival crevices of maxillary first molars on day 0 (immediately after ESP in the ibuprofen and control groups and after laser application in the laser group) and on the 1st, 3rd, and 7th days. Prior to GCF sampling, the teeth were washed, gently air-dried and isolated with cotton rolls. Standardized sterile paper strips (Periopaper, Proflow, Inc., Amityville, NY) were gently inserted into the gingival crevices until mild resistance was felt and were left in place for 30 seconds. After removing the first strip and waiting for one minute, a second strip was placed on the same side for another 30 seconds. Strips contaminated with blood or exudate were discarded. Samples were then placed separately into coded, sealed plastic microcentrifuge tubes, covered with paraffin and stored at -70 oC until the day of analysis.

ELIGIBILITY:
Inclusion Criteria:

* Being older than 18 years of age,
* Requiring ESP at the beginning of orthodontic treatment for banding of maxillary first molars,
* Intact maxillary dentition (exception of third molars),
* Fully erupted maxillary first molars without any treated or not treated apical lesions,
* Tight contacts between the posterior teeth,
* No pregnancy and lactation,
* The absence of systemic and periodontal diseases and chronic or neural pains,
* Currently not using analgesics or antibiotics that interfere the pain perception,
* No contradiction to the use of ibuprofen,
* The absence of gingival pigmentation where the laser will be applied.

Exclusion Criteria:

* Previous orthodontic treatment,
* Falling to complete the questionnaire and to continue to the follow-up appointments.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Evaluation the intensity of orthodontic pain after ibuprofen administration and laser application: levels of mediators such as interleukin 1-Beta and Substance P. | This primary outcome was evaluated trough the study completion, on average of 1 year.
  The intensity of pain observed after elastomeric separator placement was evaluated through levels of mediators such as interleukin 1-Beta and Substance P in gingival crevicular fluid objectively.
Evaluation the intensity of orthodontic pain after ibuprofen administration and laser application: visual analogue scale. | This primary outcome was evaluated trough the study completion, on average of 1 year.
  The intensity of pain observed after elastomeric separator placement was evaluated through visual analogue scale subjectively. Visual analogue scale is a 10-cm horizontal line with the number 0 representing no pain and the number 10 representing the worst pain.
Comparison of the effects of ibuprofen and laser therapy in alleviating orthodontic pain observed after elastomeric separator placement: evels of mediators such as interleukin 1-Beta and Substance P. | This primary outcome was evaluated through the study completion, on average 1 year.
  The intensity of pain observed after elastomeric separator placement was evaluated through levels of mediators such as interleukin 1-Beta and Substance P in gingival crevicular fluid objectively.
Comparison of the effects of ibuprofen and laser therapy in alleviating orthodontic pain observed after elastomeric separator placement: visual analogue scale. | This primary outcome was evaluated through the study completion, on average 1 year.
  The intensity of pain observed after elastomeric separator placement was evaluated through visual analogue scale subjectively.Visual analogue scale is a 10-cm horizontal line with the number 0 representing no pain and the number 10 representing the worst pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Van Yuzuncu Yıl University, Faculty of Dentistry, Van, Tuşba, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Krishnan V. Orthodontic pain: from causes to management--a review. Eur J Orthod. 2007 Apr;29(2):170-9. doi: 10.1093/ejo/cjl081. PMID 17488999
- [Result] Nobrega C, da Silva EM, de Macedo CR. Low-level laser therapy for treatment of pain associated with orthodontic elastomeric separator placement: a placebo-controlled randomized double-blind clinical trial. Photomed Laser Surg. 2013 Jan;31(1):10-6. doi: 10.1089/pho.2012.3338. Epub 2012 Nov 15. PMID 23153291
- [Result] Zarif Najafi H, Oshagh M, Salehi P, Babanouri N, Torkan S. Comparison of the effects of preemptive acetaminophen, ibuprofen, and meloxicam on pain after separator placement: a randomized clinical trial. Prog Orthod. 2015;16:34. doi: 10.1186/s40510-015-0104-y. Epub 2015 Oct 14. PMID 26467790
- [Result] Giannopoulou C, Dudic A, Kiliaridis S. Pain discomfort and crevicular fluid changes induced by orthodontic elastic separators in children. J Pain. 2006 May;7(5):367-76. doi: 10.1016/j.jpain.2005.12.008. PMID 16632326
- [Result] Bird SE, Williams K, Kula K. Preoperative acetaminophen vs ibuprofen for control of pain after orthodontic separator placement. Am J Orthod Dentofacial Orthop. 2007 Oct;132(4):504-10. doi: 10.1016/j.ajodo.2006.11.019. PMID 17920504
- [Result] Farias RD, Closs LQ, Miguens SA Jr. Evaluation of the use of low-level laser therapy in pain control in orthodontic patients: A randomized split-mouth clinical trial. Angle Orthod. 2016 Mar;86(2):193-8. doi: 10.2319/122214-933.1. Epub 2015 Jul 1. PMID 26132512